CLINICAL TRIAL: NCT02493179
Title: Efficacy Evaluation of the Dose Regimen of Serratiopeptidase (Serodase 5 mg Tablet) in the Treatment of Inflammation After Third Molar Surgery
Brief Title: Efficacy Evaluation of the (Serodase 5 mg Tablet) in the Treatment of Inflammation After Third Molar Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hayat Pharmaceutical Co. PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ser.01
Record Dates: First submitted 2015-04-06; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Trismus; Swelling; Inflammation
MeSH Terms: conditions — Trismus; Inflammation | interventions — serratiopeptidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Serodase 5 mg (Active Comparator): Serodase ( Serratiopeptidase) 5 mg
  Interventions: Drug: Serodase 5 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Serodase 5 mg — Serodase 5mg two tablets three times per day
  Other Names: Serratiopeptidase 5 mg tablets
  Arms: Serodase 5 mg
Drug: Placebo — Placebo two tablets three times per day
  Other Names: Placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the efficacy of dose regimen of serratiopeptidase (serodase 5 mg) as a prospective, randomized, parallel, double blind Placebo- controlled study.

DETAILED DESCRIPTION:
A prospective, randomized, parallel, double blind Placebo- controlled study to examine the efficacy of dose regimen of serratiopeptidase (serodase 5 mg) on 112 males and females volunteers in the treatment of inflammation after third molar surgery, comparing drug treatment vs placebo over a period of 20 weeks To assess the dose effectiveness of the dose regimen of Serodase 5 mg; the primary outcomes are trismus and swelling while inflammation is a secondary outcome.the expected duration of participants participation will be around 5 days divided into 4 visits, the time point of the measurment are (0,2,4 and 5 days).

The results are expected to assess the improvement of the maximal interincisal distance, reduction of swelling and improvment in the sensation of post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* participants presented with impacted lower wisdom tooth needs Buccaneers flap with buccal and distal bone removal.
* male or female 18-50
* participant is willing and able to give informed consent for paricipation in the study.
* Able and willing and able with all study requirments.

Exclusion Criteria:

* other oral surgical procedures during the same session except the removal of supernumerary third molars.
* female subject who is pregnant or lactating
* subjects has participated in any clinical research study within the previous 8 weeks.
* subjects on anti coagulant drugs .
* Unwilling participants to continue the study and those with abnormality of wound healing process.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Trimus by measuring the interincisal distance | 5 days
  the increase in the interincisal distance will show a positive effect on the Trismus
Swelling by using The Laskin method | 5 days
  the decrease in swelling will shows a positive effect on swelling based distances at predetermined time points .

SECONDARY OUTCOMES:
Post-operative pain | 5 days
  pain will be measured using the numerical pain scale from (0-10) after surgery.

REFERENCES:
- [Derived] Tamimi Z, Al Habashneh R, Hamad I, Al-Ghazawi M, Roqa'a AA, Kharashgeh H. Efficacy of serratiopeptidase after impacted third molar surgery: a randomized controlled clinical trial. BMC Oral Health. 2021 Mar 2;21(1):91. doi: 10.1186/s12903-021-01451-0. PMID 33653320